CLINICAL TRIAL: NCT02970383
Title: Narcotic Use After Minor Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Cassandra Mierisch, Orthopedic Surgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMR-CT-1
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Pain, Postoperative; Minor Surgical Procedures; Narcotics Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 group (Experimental): Initial prescription for 10 narcotic tabs
  Interventions: Behavioral: Initial prescription for 10 narcotic tabs
- 30 group (Active Comparator): Initial prescription for 30 narcotic tabs
  Interventions: Behavioral: Inital prescription for 30 narcotic tabs

INTERVENTIONS:
Behavioral: Initial prescription for 10 narcotic tabs — Reduced number of pills in initial prescription post-operatively
  Arms: 10 group
Behavioral: Inital prescription for 30 narcotic tabs
  Arms: 30 group

SUMMARY:
This study evaluates the effect of larger or smaller opioid prescriptions following minor surgery on the amount of narcotic used, patient reported satisfaction, refill requests, and leftover narcotic.

DETAILED DESCRIPTION:
Patients are randomized to receive prescriptions for either 10 or 30 tabs of 5 mg hydrocodone/325 mg acetaminophen following minor hand surgery. Patients are allowed to request additional medication as needed. Patients are contacted by phone 10-14 days after their surgery to answer a questionnaire regarding number of pills taken, number of refills requested, number of remaining pills, their satisfaction with their pain control and their surgery, and their opinion regarding the appropriateness of the prescription size.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing minor hand surgery by a participating surgeon within the study period

Exclusion Criteria:

* narcotic use within previous 3 months
* concurrent procedure
* acute trauma
* pregnancy
* allergy or other contraindication or intolerance to hydrocodone or acetaminophen
* post-operative complications
* inability to provide personal consent to the procedure or the research

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Narcotic used | 10-14 days post-op
  number of narcotic tabs taken by patient (5mg hydrocodone/325 mg acetaminophen)

SECONDARY OUTCOMES:
Number of refills requested | 10-14 days post-op
  number of times patient requested additional pain medication
Number of left over tabs | 10-14 days post-op
  Number of left over usable narcotic tabs remaining in patient possession
Patient reported efficacy of pain control | 10-14 days post-op
Patient reported satisfaction with pain control | 10-14 days post-op
Patient reported satisfaction with overall surgical experience | 10-14 days post-op
Patient Opinion Regarding Appropriateness of Size of Initial Prescription | 10-14 days post-op

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Mierisch, MD, Principal Investigator — Carilion Clinic

IPD SHARING:
Plan to Share IPD: No
none currently

REFERENCES:
- [Derived] Gaddis A, Dowlati E, Apel PJ, Bravo CJ, Dancea HC, Hagan HJ, Mierisch CM, Metzger TA, Mierisch C. Effect of Prescription Size on Opioid Use and Patient Satisfaction After Minor Hand Surgery: A Randomized Clinical Trial. Ann Surg. 2019 Dec;270(6):976-982. doi: 10.1097/SLA.0000000000003127. PMID 31730554